CLINICAL TRIAL: NCT01285284
Title: The Effect of Music Over the Tolerance to Colonoscopy ¿Does it Reduce the Discomfort, the Anxiety and the Need of Sedation? Multicentric Randomized Controlled Trial.
Brief Title: Effect of Music Over the Tolerance to Colonoscopy.
Acronym: EMOC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Clínica UC San Carlos de Apoquindo. (Unknown); Hospital Provicial Dr. Rafael Avaria Valenzuela (Unknown)
Responsible Party: Carlos Benítez Gajardo, Gastroenterology Department, Hospital Clínico de la Pontificia Universidad Católica de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-237
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-03

CONDITIONS: Pain; Anxiety
Keywords: Colonoscopy; Music; Tolerance; Pain; Anxiety; Dose of sedative drugs administered during the procedure
MeSH Terms: conditions — Pain; Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Music (Experimental): A previously defined list of songs will be administered by headphones to these patients during the colonoscopy.
  Interventions: Other: Music
- Control (Sham Comparator): These patients will receive an MP3 device (and headphones) which will be functioning but without volume.
  Interventions: Other: No music

INTERVENTIONS:
Other: Music — A previously defined list of songs will be administered by headphones to these patients.
  Arms: Music
Other: No music — No music will be administered by the headphones connected to the MP3 device.
  Arms: Control

SUMMARY:
This study will evaluate the efficacy of music (a very well selected list of songs)on improving the tolerance to the colonoscopy. The patients will be randomly assigned to receive music or not. The authors hypothesis is that music is able to improve the tolerance to colonoscopy evaluated as a reduction on the level of anxiety, on the intensity of pain experimented during the procedure and a reduction of the administered dose of midazolam during the colonoscopy.

DETAILED DESCRIPTION:
To select the music that will be administered on this trial we will performed as the first part of the study, a two fase pilot study. In the first part, five song belonging to different musical styles (Rock, Bosa Nova, Classical Music, Popular chilean music and New age) will be heard by 40 persons and the main emotion produced by every song will be registered (chosen among a previously defined list of emotions) and then rated using a visual analog scale. Thus, we will be able to select the musical style that with more frequency produce "tranquility and/or peace". Once this musical style will be selected we generate a set of songs belonging to this style. This set of songs will be validated using again a similar methodology in the second part of the pilot study to be sure that is able to produce the same emotion that the song previously evaluated. The validated set of songs will be the music that will be administered to the patients participating on a multicentric randomized controlled trial where the effect of the selected music over the tolerance to colonoscopy will be evaluated measuring the level of anxiety, the administered dose of midazolam and the intensity of pain experimented during the procedure among another variables on the experimental and the control groups, including 150 patients on each arm.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years)
* Diagnostic colonoscopy
* Signed informed consent

Exclusion Criteria:

* Hypoacusia
* Significant cognitive impairment
* Hypotension
* Signs of digestive haemorrhage (other than a small amount of rectorrhagia)
* More than moderate intensity of pain before the colonoscopy.
* Previous colorectal surgery
* allergy to midazolam or pethidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-09 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
The administered dose of midazolam | After colonoscopy is finished.
  The accumulated dose of midazolam administered during the procedure will be registered and compared between both arms.
Level of anxiety | rigth before colonoscopy and after it at the moment of discharge
  We will use a self-adminsitered questonary (STAI)

SECONDARY OUTCOMES:
Evolution of vital signs | Rigth before and during the colonoscopy
  Heart rate and blood pressure will be measured right before the colonoscopy, five and ten minutes after its start.
Colonoscopy time | During the colonoscopy
  The time elapsed since the beginning of the colonoscopy until its end.
Patient's global evaluation of the procedure | after the colonoscopy at the moment of discharge.
  After the procedure the patient will evaluate the procedure as : a)Very Bad, b)Bad, c)Good, d)Very Good.
Time since the beginning of the procedure until the discharge | since the beginning of the procedure until the discharge.
  The time elapsed since the beginning of the procedure until the discharge.
How difficult the colonoscopy was? | After the procedure.
  At the end of the colonoscopy the endocopist will be asking about how difficult the procedure was, choosing one of the following alternatives: a)Less than usual, b) as usual, c) more than usual, d) much more than usual.
Adverse effects | Since the begining of the procedure until the discharge.
  Every unexpected and adverse effect will be registered.
The level of pain | After colonoscopy at the moment of discharge
  Using a Visual Analog Scale, the intensity of pain experimented during the colonoscopy will be evaluated after the procedure on both arms.
Willing of repeating the procedure. | After colonoscopy at the moment of discharge
  After the procedure the patient will be asked about the willingness of repeating the procedure if necesary, choosing one of the following ones: a) Absolutely no, b) Possibly no, c) Possibly yes, d) Absolutely yes.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E Benítez, M.D., Principal Investigator — Gastroenterology Department. Pontificia Universidad Católica de Chile
Locations (4):
- Chile (4):
  - Hospital Provicial Dr. Rafael Avaria Valenzuela, Curanilahue, Región del Biobío
  - Centro Médico UC San Joaquín, Santiago, RM
  - Hospital Clínico. Pontificia Universidad Católica de Chile, Santiago, RM
  - Clínica UC San Carlos de Apoquindo, Santiago, Santiago Metropolitan

REFERENCES:
- [Background] Leung FW. Methods of reducing discomfort during colonoscopy. Dig Dis Sci. 2008 Jun;53(6):1462-7. doi: 10.1007/s10620-007-0025-9. PMID 17999189
- [Background] Costa A, Montalbano LM, Orlando A, Ingoglia C, Linea C, Giunta M, Mancuso A, Mocciaro F, Bellingardo R, Tine F, D'Amico G. Music for colonoscopy: A single-blind randomized controlled trial. Dig Liver Dis. 2010 Dec;42(12):871-6. doi: 10.1016/j.dld.2010.03.016. Epub 2010 May 7. PMID 20452299
- [Background] Bechtold ML, Perez RA, Puli SR, Marshall JB. Effect of music on patients undergoing outpatient colonoscopy. World J Gastroenterol. 2006 Dec 7;12(45):7309-12. doi: 10.3748/wjg.v12.i45.7309. PMID 17143946
- [Background] Harikumar R, Raj M, Paul A, Harish K, Kumar SK, Sandesh K, Asharaf S, Thomas V. Listening to music decreases need for sedative medication during colonoscopy: a randomized, controlled trial. Indian J Gastroenterol. 2006 Jan-Feb;25(1):3-5. PMID 16567885
- [Background] Ovayolu N, Ucan O, Pehlivan S, Pehlivan Y, Buyukhatipoglu H, Savas MC, Gulsen MT. Listening to Turkish classical music decreases patients' anxiety, pain, dissatisfaction and the dose of sedative and analgesic drugs during colonoscopy: a prospective randomized controlled trial. World J Gastroenterol. 2006 Dec 14;12(46):7532-6. doi: 10.3748/wjg.v12.i46.7532. PMID 17167846
- [Background] Tam WW, Wong EL, Twinn SF. Effect of music on procedure time and sedation during colonoscopy: a meta-analysis. World J Gastroenterol. 2008 Sep 14;14(34):5336-43. doi: 10.3748/wjg.14.5336. PMID 18785289
- [Background] Bechtold ML, Puli SR, Othman MO, Bartalos CR, Marshall JB, Roy PK. Effect of music on patients undergoing colonoscopy: a meta-analysis of randomized controlled trials. Dig Dis Sci. 2009 Jan;54(1):19-24. doi: 10.1007/s10620-008-0312-0. Epub 2008 May 16. PMID 18483858
- [Background] Rudin D, Kiss A, Wetz RV, Sottile VM. Music in the endoscopy suite: a meta-analysis of randomized controlled studies. Endoscopy. 2007 Jun;39(6):507-10. doi: 10.1055/s-2007-966362. PMID 17554644